CLINICAL TRIAL: NCT00363818
Title: The Association Between Platelet Function and Endothelial Function of the Brachial Artery in Healthy Subjects and in Patients With Coronary Artery Disease
Brief Title: The Association of Platelet Function and Endothelial Function of the Brachial Artery
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Michael Shechter, MD, Shlomi Matetzky, MD, PIs, Heart Institute, Sheba Medical Center
Other Study IDs: SHEBA-05-3919-MS-CTIL
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease; Endothelial Function; Thrombosis
Keywords: Endothelial function; Platelet function; Coronary artery disease; Thrombosis; Aggregation
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed study is a prospective one, and will be held on consecutive individuals undergoing the non-invasive brachial artery flow-mediated dilation (FMD) ultrasound for endothelial function at the endothelial function laboratory of the Sheba Medical Center. The study group will be divided into healthy subjects group and coronary artery disease (CAD) patients group, both of which will be analyzed in respect to age, cardiovascular risk factors and the results of the platelet and endothelial functions tests. The association between platelet and endothelial functions will be then assessed in the healthy subjects group and in the CAD patients group.

DETAILED DESCRIPTION:
Background: Previous studies have shown a significant association between endothelial dysfunction and CAD and cardiovascular risk factors. Since the endothelium is a systemic organ, endothelial dysfunction is a systemic vascular disorder which bring about a reduction in nitric oxide (NO) bioavailability accounting for distraction of the platelet function. Thus, we expect to find an association between platelet function and endothelial function assessed by the brachial artery FMD in healthy subjects and in CAD patients. Moreover, as platelet function, normally blocked by an effective anti-thrombotic therapy, is linked to the progression of atherosclerosis which, by itself is an influential process on endothelial function, we expect to find an association between endothelial function and the success of anti-thrombotic therapy.

Aim: To determine the association between platelet function and endothelial function assessed by brachial artery FMD in healthy subjects and in CAD patients, and to determine the association between anti-thrombotic therapy and endothelial function.

Methods: The proposed study is a prospective one, and will be held on consecutive individuals undergoing the non-invasive brachial artery flow-mediated dilation (FMD) ultrasound for endothelial function at the endothelial function laboratory of the Sheba Medical Center. The study group will be divided into healthy subjects group and coronary artery disease (CAD) patients group, both of which will be analyzed in respect to age, cardiovascular risk factors and the results of the platelet and endothelial functions tests. The association between platelet and endothelial functions will be then assessed in the healthy subjects group and in the CAD patients group.

The assessment of endothelial function is relatively simple and non-invasive method of short duration. Implementing this simple method to comprehend the platelet function will enable clinicians to better monitor and control the platelet inhibition in healthy subjects (for primary prevention) and in CAD patients (for secondary prevention). In addition, the FMD method can be useful in the evaluation of the success of the (antithrombocytic) treatment, the prognosis and the risk-stratification in hospitalized patients with acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (i.e., subjects without any history of chest pain or myocardial infarction, coronary artery bypass grafting surgery, coronary angiography with angioplasty and/or stenting, cerebrovascular accident, or peripheral vascular disease) with normal electrocardiograms and echocardiography on admission, and patients with coronary artery disease(i.e, patients with history of myocardial infarction, coronary artery bypass grafting operation, coronary angiography with angioplasty or stenting, heart failure secondary to coronary artery disease, or cerebrovascular accident).

Exclusion Criteria:

* Exclusion criteria included atrial fibrillation, sinus bradycardia (heart rate < 50 bpm) without pacemaker, sick sinus syndrome, second or third degree AV block, intolerance to nitrates, renal failure with serum creatinine > 3 mg/dl, history of drug or alcohol abuse, chronic liver disease, or refusal to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Heart Institute Coronary care Unit and outpatient clinic
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shechter, MD, MA, Principal Investigator — Sheba Medical Center; Shlomi Matetzky, MD, Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - Heart Center, Sheba Medical Center, Tel Litwinsky
  - The Heart Institute, Sheba Medical Center, Tel Litwinsky